CLINICAL TRIAL: NCT00495612
Title: A Phase IV, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of the Efficacy of Omalizumab in Preventing Bronchoconstriction Following Environmental Cat Dander Exposure in Patients With Cat Dander-induced Asthma
Brief Title: A Study of Omalizumab in Preventing Bronchoconstriction Following Environmental Cat Dander Exposure in Patients With Cat Dander-induced Asthma
Acronym: AERO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q4229n
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Xolair; Allergic asthma; Cat allergy
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Omalizumab (Experimental): Patients received omalizumab via subcutaneous injection either every 2 weeks or every 4 weeks for 16 weeks. The dose administered and the dosing interval were determined by serum total IgE level and body weight (measured before the start of treatment) per the study drug dosing table.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): Patients received placebo as a subcutaneous injection either every 2 weeks or every 4 weeks for 16 weeks. Patients received injections at the same time intervals as the omalizumab group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab was supplied as a sterile, white, preservative-free, lyophilized powder in single-use vials that was reconstituted with sterile water for injection.
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Placebo contained the same ingredients as the omalizumab formulation, excluding omalizumab.
  Arms: Placebo

SUMMARY:
This was a 3-center, randomized, double-blind, parallel-group, placebo-controlled study with a 16-week treatment phase to determine whether subcutaneous omalizumab, compared with placebo, reduces the degree of bronchoconstriction induced by environmental cat dander exposure in patients 18-65 years old with stable, moderate asthma and a history of cat dander-induced asthma symptoms.

DETAILED DESCRIPTION:
A cat dander allergen challenge model was used to collect data for all of the Outcome Measures. The cat allergen levels in the model are similar to those found in homes with cats and are capable of inducing lower- and upper-airway responses that have been used to assess the efficacy of several asthma and allergy therapies.

Cat allergen exposure was performed in a room furnished with upholstered furniture, a blanket, and a cat litter box. The door was kept closed at all times, except when personnel or study patients were entering or leaving the room. The ventilation system was operating at all times except during cat allergen challenges. Two neutered adult cats were kept in the room at all times and were free to move about except during challenges, at which time they are placed in wire cages. Immediately before a challenge, the blanket was shaken vigorously to distribute cat allergen throughout the room.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* 18 to 65 years of age and in general good health.
* History of moderate asthma, defined by the need for routine inhaled corticosteroids for at least the last 90 days prior to screening as well as the routine use of additional medication(s) (eg, short- or long-acting β2-agonists, leukotriene antagonist, or theophylline) to control asthma symptoms.
* History of cat dander-induced asthma in the 3 years prior to randomization.
* Cat exposure at the time of screening must remain constant throughout the duration of the study (eg, patients having cat exposure at home must continue to have regular exposure during the study; patients having no cat exposure at home must continue having no exposure at home during the study).
* Positive skin test to cat allergen, defined as a ≥ 5 mm wheal over the saline control wheal.
* Baseline forced expiratory volume in 1 second (FEV1) ≥ 70% predicted after withholding long-acting β2-agonists for > 36 hours and short-acting β2-agonists for > 6 hours.
* Eligibility per the study drug dosing table (serum IgE level ≥ 30 to ≤ 700 IU/mL and body weight ≥ 30 to ≤ 150 kg) and ability to be dosed per the dosing table.
* Less than 10 pack-years of smoking history.
* Demonstrated ≥ 20% fall in FEV1 during up to 1 hour of exposure in the cat environmental exposure chamber and ability to withstand exposure for at least 20 minutes.

Exclusion Criteria:

* Unstable asthma (defined as a hospitalization within the prior 6 months or an exacerbation requiring oral corticosteroids within 4 weeks of study entry).
* Life-threatening episode of asthma in the previous year.
* History of severe allergic reactions to cat exposure.
* Having undergone cat immunotherapy within 6 months prior to screening.
* Upper respiratory infection within 2 weeks of study entry.
* Active lung disease other than asthma.
* Significant medical illness other than asthma, including malignancies, parasitic infections, immune system disorders, and thrombocytopenia.
* History of hypersensitivity to the study drug or to drugs with similar chemical structures or to any ingredients, including excipients of the study medication or drugs related to omalizumab (eg, monoclonal antibodies, polyclonal gamma globulin).
* Documented medical history of anaphylaxis.
* Receipt of other investigational drugs within 30 days or 5 half-lives prior to screening, whichever is longer.
* Pregnant women and nursing mothers.
* Treatment with omalizumab within 12 months prior to screening.
* History of drug or alcohol abuse that, in the judgment of the investigator, may put the patient at risk for being unable to participate fully in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Solari, MD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 36 | 33
Completed | 32 | 33
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject's Decision to Withdraw | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (10.5) | 38.5 (12.3) | 36.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Percent Change in Forced Expiratory Volume in 1 Second (FEV1) Over a 1-hour Cat Allergen Exposure From Pre-challenge at Week 16
Description: Spirometry was performed prior to chamber exposure, approximately every 10 minutes during exposure, and approximately every 20 minutes after exposure until FEV1 returned to within 10% of the baseline value. A smaller change in FEV1 indicates a reduced response to the allergen exposure.
Time Frame: Week 16
Population: Modified intent-to-treat population: All randomized patients that received at least 1 dose of study drug and who had at least 1 primary efficacy data point, ie, at least 1 FEV1 measurement during the 1-hour cat allergen exposure at Week 16.
Measure: Mean (Standard Deviation); unit: Percent change from pre-challenge*hours
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 32 | 33
Percent change from pre-challenge*hours | 15.03 (15.90) | 27.80 (15.28)

2. Secondary Outcome: Percent Change in Forced Expiratory Volume in 1 Second (FEV1) at 20 Minutes of a 1-hour Cat Allergen Exposure From Pre-challenge at Week 16
Description: Spirometry was performed prior to chamber exposure, approximately every 10 minutes during exposure, and approximately every 20 minutes after exposure until FEV1 returned to within 10% of baseline value. A smaller change in FEV1 indicates a reduced response to the allergen exposure.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 32 | 33
Percent change | 15.28 (18.00) | 29.97 (17.77)

3. Secondary Outcome: Maximum Percent Change in Forced Expiratory Volume in 1 Second (FEV1) During a 1-hour Cat Allergen Exposure From Pre-challenge at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 32 | 33
Percent change | 21.07 (17.68) | 33.52 (16.03)

4. Secondary Outcome: Area Under the Curve (AUC) of Change in Chest Symptom Score During a 1-hour Cat Allergen Exposure From Pre-challenge at Week 16
Description: The chest symptom score was defined as the total of 4 sub-scores: Chest tightness, wheezing, shortness of breath, and cough. Each sub-score was rated by the patient on a scale of 0-3 (0=none, 1=mild, 2=moderate, and 3=severe) immediately prior to and approximately every 5 minutes during chamber exposure. The maximum chest symptom score was 12 points. A lower score indicates a reduced response to the allergen exposure and fewer respiratory symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 32 | 33
Units on a scale*hours | 2.205 (2.066) | 5.602 (2.873)

5. Secondary Outcome: Area Under the Curve (AUC) of Change in Nasal-ocular Symptom Score (NOSS) During a 1-hour Cat Allergen Exposure From Pre-challenge at Week 16
Description: The NOSS was defined as the total of 4 sub-scores: Nasal congestion, rhinorrhea, nasal pruritus, ocular pruritus, and ocular tearing. Each sub-score was rated by the patient on a scale of 0-3 (0=none, 1=mild, 2=moderate, and 3=severe) immediately prior to and approximately every 5 minutes during chamber exposure. The maximum NOSS was 15 points. A lower score indicates a reduced response to the allergen exposure and fewer nasal-ocular symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 32 | 33
Units on a scale*hours | 2.448 (1.720) | 5.192 (3.141)

6. Secondary Outcome: Duration of Allergen Exposure During the Cat Allergen Exposure Challenge at Week 16
Description: The challenge was stopped if a patient stated that they were extremely uncomfortable and would like to leave the room, the FEV1 has decreased by 50% from the baseline value, or after 60 minutes of exposure. The duration of allergen exposure was the time from when the patient entered the exposure room until the challenge stopped, with a maximum of 60 minutes. A longer duration indicates greater tolerance of the allergen exposure.
Time Frame: Week 16
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 32 | 33
Minutes | 50 [37 to NA] — The upper limit of the confidence interval could not be estimated due to too few events, defined as exiting the challenge before 60 minutes. | 22 [10 to 30]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time informed consent was given until a patient completed the study or discontinued prematurely.
Description: Safety analyses were based on the treated subjects. Treated subjects were defined as randomized subjects who received at least 1 dose of study drug. The treatment groups were based on the treatment subjects actually received regardless of their assigned treatment.
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/33
Other Adverse Events (participants affected / at risk) | 26/36 | 31/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=36) | Placebo (N=33)
Nausea (Gastrointestinal disorders) | 0 | 2
Chest discomfort (General disorders) | 2 | 1
Hypersensitivity (Immune system disorders) | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 5 | 5
Urinary tract infection (Infections and infestations) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 7 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.